CLINICAL TRIAL: NCT07191158
Title: Evaluation of Three-Dimensional Printed Orthodontic Molar Distalizer (Randomized Clinical Trial)
Brief Title: Evaluation of Three-Dimensional Printed Orthodontic Molar Distalizer
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mushriq F. Abid, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1020425
Record Dates: First submitted 2025-08-29; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Tooth Movement Techniques; Distalization by Miniscrews
Keywords: Distalization; tooth movement; 3D printing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be a single blinded because both the patients and the investigator will be aware of the allocation during treatment, but the cephalograms and digital models will be scored and coded by an independent person, i.e. pre-and post-treatment cephalograms and digital models will be analyzed after replacing the patients' names with codes, and the examiner conducting the measurement analysis will be unaware of the group to which the patient has been allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 distalization (Active Comparator): Conventional miniscrew-supported distal jet appliance
  Interventions: Device: Group 1 conventional
- Group 2 (interventional) (Experimental): New 3D printed miniscrew-supported molar distalizers
  Interventions: Device: Group 2 3D printed

INTERVENTIONS:
Device: Group 1 conventional — Conventional miniscrew-supported distal jet appliance
  Arms: Group 1 distalization
Device: Group 2 3D printed — New 3D printed miniscrew-supported molar distalizers
  Arms: Group 2 (interventional)

SUMMARY:
A randomized clinical trial to evaluate a newly designed 3D printed miniscrew-supported molar distalization device in comparison to the conventional miniscrew-supported distal jet appliance in correction of Class II malocclusion and upper arch crowding.

DETAILED DESCRIPTION:
It is a multicenter randomized clinical trial with two parallel arms. The patients will be randomly divided into two groups, group one: conventional miniscrew-supported distal jet appliance will be used while for group two, new 3D printed miniscrew-supported molar distalizers is going to be utilized. Lateral cephalometric x-ray and digital models of upper arch will be taken before starting the treatment (T0) and at the end of molar distalization (T1). The effectiveness of the two appliances will be assessed and measured comparing patient's records before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Class II molar relationships bilaterally, with fully erupted 2nd molar.
2. No or minor crowding on the mandible to [reserve Class I posterior occlusion after treatment.
3. Good oral health free from caries and periodontal problems at the start of treatment.

   -

Exclusion Criteria:

1. Previous history of orthopedic and/or orthodontic treatment.
2. Patients with cleft lip and palate and/or craniofacial syndrome
3. Patients with bad oral habit.
4. Active periodontal disease.
5. Sever rotation of maxillary molars. -

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The rate of molar Distalization | 6 months
  • The efficiency of molar distalization in terms of the amount of molar distalization, degree of distal tipping and bodily translation movements by using a lateral cephalogram linear and angular measurements.

SECONDARY OUTCOMES:
Patient discomfort | 10 days
  • Patient's pain and discomfort using visual analogue scale (VAS). The minimum score is zero and the maximum score is 10.
Molar distalization | 6 months
  The efficiency of molar distalization in terms of the amount of molar distalization, degree of distal tipping and bodily translation movements by using a lateral cephalogram linear and angular measurements. - The efficiency of molar distalization in terms of the amount of molar distalization, - degree of distal tipping and bodily translation movements by using a lateral cephalogram linear and angular measurements

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry-University of Baghdad, Baghdad, Al-Russafa, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cassetta M, Brandetti G, Altieri F. Miniscrew-supported distal jet versus conventional distal jet appliance: A pilot study. J Clin Exp Dent. 2019 Jul 1;11(7):e650-e658. doi: 10.4317/jced.55780. eCollection 2019 Jul. PMID 31516664